CLINICAL TRIAL: NCT07093359
Title: Double-blind Randomised Controlled Trial for Treatment of Gastro-Oesophageal Reflux Disease; LINX Management System vs. Fundoplication (GOLF)
Brief Title: LINX vs Fundoplication
Acronym: GOLF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: King's College London (Other); Imperial College London (Other); Oxford University Hospitals NHS Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other); University of Bristol (Other); University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRAS 331404; NIHR152268 (Other Grant/Funding Number: National Institute for Health and Care Research); ISRCTN 13533177 (Registry Identifier: ISRCTN: the UK's Clinical Study Registry)
Record Dates: First submitted 2025-07-02; First posted 2025-07-30 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-06

CONDITIONS: Gastro-oesophageal Reflux Disease
Keywords: LINX; GORD; GERD; Fundoplication; REFLUX; ANTI REFLUX
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laparoscopic or robotic fundoplication (Active Comparator): Participants randomised to laparoscopic or robotic fundoplication will receive surgical treatment for managing GORD including a total or partial fundic wrap behind or in front of the distal oesophagus and gastro-oesophageal junction.
  Interventions: Procedure: Laparoscopic or robotic fundoplication
- Laparoscopic or robotic LINX procedure (Experimental): Participants randomised to laparoscopic or robotic magnetic sphincter augmentation (LINX procedure) will receive surgical treatment under general anaesthesia, with placement of the LINX device around the distal oesophagus. The LINX device comprises titanium beads with magnets in the centre.
  Interventions: Procedure: Laparoscopic or robotic LINX procedure

INTERVENTIONS:
Procedure: Laparoscopic or robotic LINX procedure — Participants randomised to laparoscopic or robotic magnetic sphincter augmentation (LINX procedure) will receive surgical treatment under general anaesthesia, with placement of the LINX device around the distal oesophagus. The LINX device comprises titanium beads with magnets in the centre.
  Arms: Laparoscopic or robotic LINX procedure
Procedure: Laparoscopic or robotic fundoplication — Participants randomised to laparoscopic or robotic fundoplication will receive surgical treatment for managing GORD including a total or partial fundic wrap behind or in front of the distal oesophagus and gastro-oesophageal junction.
  Arms: Laparoscopic or robotic fundoplication

SUMMARY:
Reflux disease can severely impact upon quality-of-life and lead to complications, including ulceration of the oesophagus. It is often controlled with self-help measures and medication. However, sometimes surgery is recommended. The current standard surgical treatment is called a fundoplication. This operation is carried out through keyhole (laparoscopic) surgery, and tightens the lower oesophagus to prevent reflux. Fundoplication is very safe and improves the quality-of-life of most patients. However, many patients have gas bloating, difficulty swallowing and recurrence of their reflux symptoms. As an alternative, some surgeons use a device called LINX, using a keyhole procedure. LINX is a magnetic device that wraps around the lower oesophagus to prevent reflux. Studies suggest that LINX may cause fewer complications, with a similar improvement in quality-of-life. However, there is a need for better evidence to compare LINX with fundoplication in the surgical treatment of reflux disease. GOLF is a multi-centre study designed which to determine if LINX achieves similar reflux control and improves symptoms compared to fundoplication. GOLF measures: (1) quality of life,(2) surgical complications, including need for additional treatment, (3) financial cost-effectiveness and (4) objectively measure the presence of acid that has refluxed into the lower oesophagus. GOLF aims randomise 460 patients to receive fundoplication or the LINX device. It will be conducted across at least 16 UK and 7 European specialist surgical centres. All participants will be followed up at 6 weeks, 6, 12 and 24 months to assess which treatment offers the best results after surgery. A quality assurance programme within participating centres will ensure that procedures are completed to a high-quality standard. Study results will incorporate a patient and public involvement programme, which will inform national and international guidelines for the surgical treatment of reflux disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and above
2. Willing and able to give informed consent
3. Patients with GORD insufficiently controlled by medical therapy or intolerance to medical therapy being considered for anti-reflux surgery
4. Symptomatic and objectively defined GORD; endoscopy with appearances or biopsies consistent with reflux oesophagitis, or 24-hour pH study or BRAVO test of the oesophagus consistent with GORD
5. No hiatal hernia or hiatal hernia <5 cm in length
6. Adequate lower oesophageal motility as defined by preoperative oesophageal manometry study. Oesophageal manometry will show a mean contractile amplitude of >30 mmHg or DCI >450 mmHg-s-cm in 70% of swallows.

Exclusion Criteria:

1. Unsuitable for surgical intervention due to medical conditions precluding general anaesthesia
2. Suspected or known allergies to titanium, stainless steel, nickel, or ferrous materials
3. Previous anti-reflux or gastric surgery
4. Previous or planned neurosurgical intervention
5. Oesophageal manometry showing complete absence of lower oesophageal contractility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Symptomatic GORD and health-related quality of life (HRQL) assessed using the GORD-HRQL questionnaire | 24 months following surgery

SECONDARY OUTCOMES:
Prevalence of gas bloating measured using participant-reported outcomes/GORD-HRQL and Foregut Symptom Questionnaire | 24 months postoperatively
Prevalence of inability to belch measured using participant-reported outcomes/GORD-HRQL and Foregut Symptom Questionnaire | 24 months postoperatively
Prevalence of symptomatic GORD, inability to belch and gas bloating measured using participant-reported outcomes/GORD-HRQL and Foregut Symptom Questionnaire | 6 weeks, 6 and 12 months after surgery
Severity of dysphagia and regurgitation measured using participant-reported outcomes/GORD-HRQL questionnaire | 6 weeks, 6, 12 and 24 months postoperatively
Global HRQL measured using participant-reported outcomes/EQ-5D-5L questionnaire | 6 weeks, 6, 12 and 24 months postoperatively
Utilisation of anti-GORD medications measured using participant-reported outcomes/questionnaire | 6 weeks, 6, 12 and 24 months postoperatively
24-hour pH measurement measured using participant's medical records/24-hour pH measurement or BRAVO test | 12 months postoperatively
Postoperative complication rates, including reoperation and endoscopic reintervention, measured using participant's medical records/postoperative outcomes | 30-day, 90-day, 12 and 24-month
Cost-effectiveness of both treatments as measured by incremental cost per quality-adjusted life year (QALY) | 6 weeks, 6, 12 and 24 months postoperatively

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - Guy's and St Thomas's NHS Foundation Trust, Guy's and St Thomas's Hospital, Oxford, Oxfordshire
  - Imperial College Healthcare NHS Trust, St Mary's Hospital, Oxford, Oxfordshire
  - Leeds Teaching Hospitals NHS Trust, St James's University Hospital, Oxford, Oxfordshire
  - Oxford University Hospitals NHS Foundation Trust, Churchill Hospital, Oxford, Oxfordshire
  - University Hospital Southampton NHS Foundation Trust, Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: No
The data-sharing plans for the current study are unknown and will be made available at a later date.

REFERENCES:
- See also: Study website — https://www.nds.ox.ac.uk/research/surgical-intervention-trials-unit/golf